CLINICAL TRIAL: NCT05373472
Title: A Randomized, Double-blind, Dose-exploring, Placebo-controlled, Multi-center Phase II Clinical Trial Evaluating the Safety and Immunogenicity of COVID-19 mRNA Vaccine in Adults Aged 18 Years and Older
Brief Title: Phase II Clinical Trial of COVID-19 mRNA Vaccine in Adults Aged 18 Years and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-NCVM-002
Record Dates: First submitted 2022-05-12; First posted 2022-05-13 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
Keywords: COVID; mRNA; Vaccine; Placebo; Safety; Immunogenicity
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Vaccine Group, low dose, 18-59 year-old (Experimental): 2 doses of COVID-19 mRNA vaccine (30µg, 0.3 ml) on Day 0 and Day 21
  Interventions: Biological: COVID-19 mRNA vaccine
- Vaccine Group, low dose, 60 year-old and above (Experimental): 2 doses of COVID-19 mRNA vaccine (30µg, 0.3 ml) on Day 0 and Day 21
  Interventions: Biological: COVID-19 mRNA vaccine
- Vaccine Group, high dose, 18-59 year-old (Experimental): 2 doses of COVID-19 mRNA vaccine (50µg, 0.5 ml) on Day 0 and Day 21
  Interventions: Biological: COVID-19 mRNA vaccine
- Vaccine Group, high dose, 60 year-old and above (Experimental): 2 doses of COVID-19 mRNA vaccine (50µg, 0.5 ml) on Day 0 and Day 21
  Interventions: Biological: COVID-19 mRNA vaccine
- Placebo Group, low dose, 18-59 year-old (Placebo Comparator): 2 doses of placebo (0µg, 0.3 ml) on Day 0 and Day 21
  Interventions: Biological: Placebo
- Placebo Group, low dose, 60 year-old and above (Placebo Comparator): 2 doses of placebo (0µg, 0.3 ml) on Day 0 and Day 21
  Interventions: Biological: Placebo
- Placebo Group, high dose, 18-59 year-old (Placebo Comparator): 2 doses of placebo (0µg, 0.5 ml) on Day 0 and Day 21
  Interventions: Biological: Placebo
- Placebo Group, high dose, 60 year-old and above (Placebo Comparator): 2 doses of placebo (0µg, 0.5 ml) on Day 0 and Day 21
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: COVID-19 mRNA vaccine — 2 doses of vaccine on Day 0 and Day 21
  Arms: Vaccine Group, high dose, 18-59 year-old; Vaccine Group, high dose, 60 year-old and above; Vaccine Group, low dose, 18-59 year-old; Vaccine Group, low dose, 60 year-old and above
Biological: Placebo — 2 doses of placebo on Day 0 and Day 21
  Arms: Placebo Group, high dose, 18-59 year-old; Placebo Group, high dose, 60 year-old and above; Placebo Group, low dose, 18-59 year-old; Placebo Group, low dose, 60 year-old and above

SUMMARY:
To evaluate the safety and immunogenicity of COVID-19 mRNA vaccine in people aged 18 years and older, 300 participants will be enrolled and divided into two groups: low- and high-dose groups. Each dose group (150 people) will be divided into 2 age groups (75 each):18 to 59 years old and ≥ 60 years old. The subjects will be randomized into vaccine group or placebo group in a ratio of 2:1. Subjects will complete 2 doses of vaccination on Day 0 and Day 21, in which the low-dose group will received 0.3 ml of the study vaccine or placebo, and the high dose group received 0.5 ml of the study vaccine or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and above with BMI not lower than 18 ;
2. Volunteers are able and willing to comply with the requirements of the clinical trial protocol, and volunteers or witnesses can sign informed consent forms;
3. Willing to discuss the medical history with the investigator or doctor and allow access to all medical records related to this trial;
4. Provide 48-hour PCR negative report;
5. Have not received any other COVID-19 vaccines.

Exclusion Criteria:

* Criteria for exclusion of the first dose

  1. Other medical or psychiatric conditions, including recent (within the past year) or current presence of suicidal ideation/behavior, or laboratory abnormalities that may increase the risk of participating in the study, or subjects who are not suitable to participate in the study according to the investigator's judgment;
  2. Positive for human immunodeficiency virus (HIV);
  3. History of infection or disease history of Middle East Respiratory Syndrome (MERS), SARS or other coronaviruses or related immunizations;
  4. History of serious adverse reactions associated with the vaccine and/or a history of severe allergic reactions (e.g., anaphylaxis) to any component of the vaccine under study;
  5. Immunocompromised patients with known or suspected immunodeficiency identified by medical history and/or physical examination;
  6. Bleeding constitution or condition associated with prolonged bleeding which investigators believe that intramuscular injection is contraindicated;
  7. Women who test positive for blood pregnancy or are breastfeeding, volunteers or their partners have a pregnancy plan within 12 months;
  8. Severe hypertension and uncontrollable medication (on-site measurement: systolic blood pressure ≥ 160mmHg, diastolic blood pressure ≥ 100mmHg);
  9. Have a serious chronic disease or the condition is in the progression period can not be smoothly controlled, such as diabetes, thyroid disease, etc.;
  10. History of severe myocarditis, pericarditis and other heart diseases;
  11. Plans to receive other vaccines within 28 days before and after receiving the test vaccine;
  12. Those receiving immunosuppressive therapy, including cytotoxic drugs or systemic corticosteroids, such as for cancer or autoimmune diseases, or who were scheduled to receive treatment throughout the study period. If systemic corticosteroids are used in a short period of time (< 14 days) for the treatment of acute illness, subjects should not enter this study until at least 28 days after corticosteroid therapy has been discontinued prior to study vaccination. Inhalation/spraying, intra-articular, intraskeletal, or topical (skin or eyes) use of corticosteroids is permitted;
  13. Receiving blood/plasma products or immunoglobulins 60 days prior to study vaccination or plan to receive for the entire study duration;
  14. Engage in other interventional studies within 28 days prior to entering the study and/or during the study's participation;
  15. Participated in other interventional studies of lipid-containing nanoparticles;
  16. Have symptoms of COVID-19 such as respiratory symptoms, fever, cough, shortness of breath, and dyspnea;
  17. Fever, axillary temperature > 37.0 °C.

Second dose exclusion criteria:

1. Severe allergic reactions occur after the first vaccination;
2. Serious adverse reactions with causal relationship during the first vaccination;
3. Those who are newly discovered or newly occurring after the first vaccination do not meet the inclusion criteria of the first dose or meet the exclusion criteria of the first dose, and the investigator shall decide whether to continue to participate in the study;
4. Other reasons for exclusion that the investigators believe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of wild type neutralizing antibodies | 28 days after complete immunization
  GMT of wild type neutralizing antibodies
Immunogenicity of wild type neutralizing antibodies | 28 days after complete immunization
  Sero-conversation rate of wild type neutralizing antibodies
The incidence of adverse reactions (AR) | Within 14 days of each vaccination
  To evaluate the incidence of adverse reactions (AR) in all subjects

SECONDARY OUTCOMES:
The incidence of adverse reactions (AR) | Within 28 days of complete immunization
  To evaluate the incidence of adverse reactions (AR) in all subjects
The incidence of adverse reactions (AR) | Within 60 minutes of each vaccination
  To evaluate the incidence of adverse reactions (AR) in all subjects
The incidence of SAE, MAE and AESI | 12 months after complete vaccination
  To evaluation the incidence of SAE, MAE, and AESI in all subjects
Immunogenicity of wild type neutralizing antibodies | Before the 1st dose, 14 days after the 2nd dose, and 3, 6, 12 months after the 2nd dose
  Sero-conversation rate of wild type neutralizing antibodies
Immunogenicity of wild type neutralizing antibodies | Before the 1st dose, 14 days after the 2nd dose, and 3, 6, 12 months after the 2nd dose
  GMT of wild type neutralizing antibodies
Immunogenicity of wild type neutralizing antibodies | Before the 1st dose, 14 days after the 2nd dose, and 3, 6, 12 months after the 2nd dose
  GMI of wild type neutralizing antibodies
Immunogenicity of wild type neutralizing antibodies | 28 days after complete immunization
  GMI of wild type neutralizing antibodies
Immunogenicity of anti-S-RBD Ig G antibodies | Before the 1st dose, 14 days after the 2nd dose, 28 days after the 2nd dose and month 3,6,12 months after 2nd vaccination
  Sero-conversation rate of anti-S-RBD Ig G antibodies
Immunogenicity of anti-S-RBD Ig G antibodies | before the 1st dose, 14 days after the 2nd dose, 28 days after the 2nd dose and month 3,6,12 months after 2nd vaccination
  GMC of anti-S-RBD Ig G antibodies
Immunogenicity of anti-S-RBD Ig G antibodies | before the 1st dose, 14 days after the 2nd dose, 28 days after the 2nd dose and month 3,6,12 months after 2nd vaccination
  GMI of anti-S-RBD Ig G antibodies
Cellular immunity | Before the 1st dose, 14 days after the 2nd dose, 28 days after the 2nd dose and month 3,6,12 months after 2nd vaccination
  The response levels and positive rates of IL-2 produced by S protein RBD by ICS in the first 15 subjects in each group
Cellular immunity | Before the 1st dose, 14 days after the 2nd dose, 28 days after the 2nd dose and month 3,6,12 months after 2nd vaccination
  The response levels and positive rates of IL-4 produced by S protein RBD by ICS in the first 15 subjects in each group
Cellular immunity | Before the 1st dose, 14 days after the 2nd dose, 28 days after the 2nd dose and month 3,6,12 months after 2nd vaccination
  The response levels and positive rates of IL-5 produced by S protein RBD by ICS in the first 15 subjects in each group
Cellular immunity | Before the 1st dose, 14 days after the 2nd dose, 28 days after the 2nd dose and month 3,6,12 months after 2nd vaccination
  The response levels and positive rates of IL-17 produced by S protein RBD by ICS in the first 15 subjects in each group
Cellular immunity | Before the 1st dose, 14 days after the 2nd dose, 28 days after the 2nd dose and month 3,6,12 months after 2nd vaccination
  The response levels and positive rates of IFN-γ produced by S protein RBD by ICS in the first 15 subjects in each group
Changes in laboratory indicators | Before 1st dose and 28 days after second dose
  Changes in white blood cell count
Changes in laboratory indicators | Before 1st dose and 28 days after second dose
  Changes in neutrophils
Changes in laboratory indicators | Before 1st dose and 28 days after second dose
  Changes in lymphocyte count
Changes in laboratory indicators | Before 1st dose and 28 days after second dose
  Changes in platelet count
VOC/VOI serum cross neutralization | 28 days after complete immunization
  To evaluated the level of VOC/VOI serum cross neutralization results in all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Dong, Principal Investigator — Beijing Friendship Hospital; Kexin Zhao, Principal Investigator — Hebei Petro China Center Hospital; Tao Huang, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (3):
- China (3):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Hebei Petro China Center Hospital, Langfang, Hebei
  - Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan

REFERENCES:
- [Derived] Jin Z, Wu J, Huang T, Zhao K, Zhang M, Liu J, Song J, Yin H, Wu X, Liu J, Zhu T, Huang H, Li J, Wang H, Gou J, Dong R. Safety, immunogenicity, persistence and dose evaluation of the CS-2034 mRNA COVID-19 vaccine: a phase II randomized controlled trial in healthy Chinese adults. BMC Infect Dis. 2025 Nov 20;25(1):1625. doi: 10.1186/s12879-025-12053-4. PMID 41267026